CLINICAL TRIAL: NCT00193479
Title: A Phase II Trial of Brief Duration Combination Chemotherapy and Rituximab With Prophylactic Pegfilgrastim, Followed by Maintenance Rituximab, in Elderly/Poor Performance Status Patients With Large B-Cell Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy and Rituximab With Pegfilgrastim Followed by Rituximab, in Large B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LYM 28
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; Mitoxantrone; Vincristine; Prednisone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyclophosphamide/Vincristine/Rituximab +/- Mitoxantrone (Experimental): All patients receive three courses of combination chemotherapy/rituximab followed by pegfilgrastim, administered at 21-day intervals. Treatment administered is as follows: cyclophosphamide 500mg/m2 IV day 1; mitoxantrone 10mg/m2 IV day 1; vincristine 1.0mg/m2 (maximum 2mg) IV day 1; prednisone 80mg PO days 1 - 5; rituximab 375mg/m2 IV day 1.
  Interventions: Drug: Cyclophosphamide; Drug: Mitoxantrone; Drug: Vincristine; Drug: Prednisone; Drug: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide
  Other Names: Cytoxan
Drug: Mitoxantrone — Mitoxantrone
  Other Names: Novantrone
Drug: Vincristine — Vincristine
  Other Names: Oncovin
Drug: Prednisone — Prednisone
Drug: Rituximab — Rituximab
  Other Names: Rituxan

SUMMARY:
The purposes of this trial are to decrease toxicity and improve treatment effectiveness elderly patients. With a short course of chemotherapy with cyclophosphamide, mitoxantrone, vincristine, and prednisone with concurrent administration of rituximab it is likely to be as effective as longer programs, and will certainly be better tolerated by this patient group. The addition of maintenance therapy may result in substantial prolongation of remission duration.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will receive:

* Cyclophosphamide + Mitoxantrone + Vincristine + Prednisone + Rituximab

Patients that are not considered candidates for anthracycline therapy will not receive mitoxantrone. Patients with objective response (partial or complete response) or stable disease will receive Rituximab maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Histologically documented large B-cell, CD20-positive non-Hodgkin's lymphoma
* No previous treatment
* Clinical stage II, III, or IV by the Ann Arbor Staging Criteria
* Age > 70 years
* ECOG performance status 0, 1, or 2
* Adequate bone marrow, liver and kidney function
* Must give written informed consent prior to entering this trial

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Age < 18 years
* Central nervous system involvement with lymphoma
* Coexistent active malignancies treated within five years
* Active infection precluding the use of combination chemotherapy
* HIV infection
* Pregnant or lactating

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-04; Primary Completion 2008-07 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (2):
- United States (2):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Tennessee Oncology, Nashville, Tennessee

REFERENCES:
- [Result] Hainsworth JD, Flinn IW, Spigel DR, Clark BL, Griner PL, Vazquez ER, Doss HH, Shipley D, Franco LA, Burris HA 3rd, Greco FA; Sarah Cannon Oncology Research Consortium. Brief-duration rituximab/chemotherapy followed by maintenance rituximab in patients with diffuse large B-cell lymphoma who are poor candidates for R-CHOP chemotherapy: a phase II trial of the Sarah Cannon Oncology Research Consortium. Clin Lymphoma Myeloma Leuk. 2010 Feb;10(1):44-50. doi: 10.3816/CLML.2010.n.004. PMID 20223728
- See also: Published article in Clinical Lymphoma, Myeloma and Leukemia — http://cigjournals.metapress.com/content/418721241w307702/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-eight of 51 patients (94%) completed the initial three courses of rituximab/chemotherapy. Forty-four of the 48 patients (92%) received the Rituximab maintenance therapy.
Groups:
- CNOP (CVP)/Rituximab/Pegfilgrastim Followed by Rituximab: Cyclophosphamide 500mg/m2 IV day 1; Mitoxantrone 10mg/m2 IV day 1; Vincristine 1.0mg/m2 IV day 1; Prednisone 80mg PO days 1-5; Rituximab 375mg/m2 IV day 1; Pegfilgrastim 6mg SQ, day 2 OR Cyclophosphamide 500mg/m2 IV day 1; Vincristine 1.0mg/m2 IV day 1; Prednisone 80mg PO days 1-5; Rituximab 375mg/m2 IV day 1; Pegfilgrastim 6mg SQ, day 2
Period: Induction Chemotherapy
Arm/Group | CNOP (CVP)/Rituximab/Pegfilgrastim Followed by Rituximab
Started | 51
Completed | 48
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Disease Progression | 1
Period: Maintenance Rituximab
Arm/Group | CNOP (CVP)/Rituximab/Pegfilgrastim Followed by Rituximab
Started | 48
Completed | 44
Not Completed | 4
Not completed — Opted for full course rituximab/chemotherapy | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | CNOP (CVP)/Rituximab/Pegfilgrastim Followed by Rituximab
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 78 [61 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 Months
Measure: Number; unit: percentage of patients
Arm/Group | CNOP (CVP)/Rituximab/Pegfilgrastim Followed by Rituximab
Number analyzed (Participants) | 48
percentage of patients | 81

ADVERSE EVENTS:
Arm/Group | CNOP (CVP)/Rituximab/Pegfilgrastim Followed by Rituximab
Serious Adverse Events (participants affected / at risk) | 24/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNOP (CVP)/Rituximab/Pegfilgrastim Followed by Rituximab (N=51)
Pneumonia (Infections and infestations) | 2 (2)
Perforated colon (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
CVA (Nervous system disorders) | 4 (4)
Infection of bilateral heel ulcer wounds (Infections and infestations) | 1 (1)
Infection, L ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Concussion, related to fall (Nervous system disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fractured hip (Musculoskeletal and connective tissue disorders) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Fractured ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
CHF (Cardiac disorders) | 1 (1)
Acute chronic fractures on lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Gross hematuria (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Diverticulosis (Gastrointestinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
New primary lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Acute renal failure (Skin and subcutaneous tissue disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Intractable neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right lower thigh pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Intramedullary spinal cord mass (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNOP (CVP)/Rituximab/Pegfilgrastim Followed by Rituximab (N=51)
Alopecia (Skin and subcutaneous tissue disorders) | 30 (152)
Anemia (Blood and lymphatic system disorders) | 35 (169)
Anorexia (Gastrointestinal disorders) | 29 (85)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (42)
Cardiac Toxicity (Cardiac disorders) | 8 (17)
Chills/Rigor (General disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 21 (47)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 12 (19)
Dizziness (Nervous system disorders) | 8 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema (General disorders) | 8 (18)
Fatigue (General disorders) | 44 (305)
Fever (General disorders) | 8 (12)
Headache (Nervous system disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (21)
Hypertension (Cardiac disorders) | 4 (4)
Hypotension (Cardiac disorders) | 4 (6)
Infection (Infections and infestations) | 19 (36)
Insomnia (General disorders) | 6 (8)
Leukopenia (Blood and lymphatic system disorders) | 25 (82)
Mucositis (Gastrointestinal disorders) | 5 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (26)
Nausea (Gastrointestinal disorders) | 18 (31)
Neuropathy (Nervous system disorders) | 4 (6)
Neutropenia (Blood and lymphatic system disorders) | 21 (54)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 7 (29)
Rash/Skin Irritation (Skin and subcutaneous tissue disorders) | 8 (20)
Stomatitis (Gastrointestinal disorders) | 6 (8)
Taste Alteration (Gastrointestinal disorders) | 3 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (59)
Vomiting (Gastrointestinal disorders) | 9 (13)
Weakness (General disorders) | 13 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.